CLINICAL TRIAL: NCT06835803
Title: Enhanced Local Intensified Radiation Therapy in Elderly Glioblastoma (ELITE-GBM): A Phase 2 Hybrid Randomized Trial Leveraging External Data
Brief Title: Enhanced Local Intensified Radiation Therapy in Elderly Glioblastoma: A Phase 2 Hybrid Randomized Trial
Acronym: ELITE-GBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rifaquat M. Rahman, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-637
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma (GBM)
Keywords: glioblastoma; elderly glioblastoma; hypofractionation
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The study will use a hybrid design that also leverages an external control dataset in order to adjust the randomization ratio in favor of the experimental arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-escalated hypofractionated radiation over 3 weeks (Experimental)
  Interventions: Radiation: Dose-escalated radiation therapy
- Standard hypofractionated radiation over 3 weeks (Active Comparator)
  Interventions: Radiation: Standard hypofractionated radiation

INTERVENTIONS:
Radiation: Dose-escalated radiation therapy — Dose-escalated radiation therapy involves higher doses of radiation therapy each day of treatment over the three week course of radiation therapy
  Arms: Dose-escalated hypofractionated radiation over 3 weeks
Radiation: Standard hypofractionated radiation — Standard hypofractionated radiation therapy over 3 weeks
  Arms: Standard hypofractionated radiation over 3 weeks

SUMMARY:
Glioblastoma (GBM) is an aggressive malignancy of the central nervous system. Older adults with GBM have a unique constellation of medical, psychosocial, and supportive care needs. To address these challenges, prior work has evaluated the feasibility of hypofractionation, a treatment approach delivering fewer, larger radiation dosages over a shorter time period. Common hypofractionated regimens deliver a lower biologically equivalent radiation dose than the conventional regimens used for younger adults. Whether dose escalated hypofractionation can further improve outcomes in older adults remains unclear.

This will be a hybrid randomized control trial comparing the efficacy and safety of dose-escalated and standard hypofractionated radiotherapy among older adults with newly-diagnosed glioblastoma compared to standard three-week course. This research study involves the administration of radiation therapy. Radiation will either be delivered at the standard daily dose or at an increased daily dose over a three weeks course of radiation treatment.

Research study procedures will include a screening evaluation to assess eligibility, as well as clinical visits for radiation delivery and to assess symptoms during treatment and at scheduled follow-up times.

Participants will be randomly assigned to one of the two arms of the trial:

1. Standard hypofractionated radiation over 3 weeks
2. Dose-escalated hypofractionated radiation over 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of WHO grade 4 glioblastoma (IDH wild-type by immunohistochemistry or sequencing). Histopathology must be confirmed by central review.
* Newly diagnosed disease, with time elapsed from diagnostic surgery/resection <8 weeks.
* Age ≥ 65 years old at time of glioblastoma diagnosis
* Adequate functional status as measured by a ECOG Performance Status 0, 1 or 2, at time of enrollment.
* Adequate hematological, renal and hepatic functions as defined by the following required laboratory values obtained within 45 days prior to randomization:

Platelet count ≥ 100 x 10^9/L (100,000 cells/mm^3) Serum creatinine ≤ 1.5 times the upper limit of normal Total serum bilirubin ≤ 1.5 times the upper limit of normal ALT (SGPT) < 2.5 times the upper limit of normal and/or AST (SGOT) < 2.5 times the upper limit of normal

-Patient may have received corticosteroids, but must be on a stable or decreasing dose for at least 14 days prior to randomization.

Exclusion Criteria:

* Participants with recurrent glioma.
* Participants with evidence of spinal, leptomeningeal, or more distant disease.
* Participants with another active central nervous system malignancies requiring treatment.
* Participants with a second invasive malignancy that is A) incompletely treated or requiring ongoing treatment, or B) reasonably anticipated to be associated with a median overall survival of less than 1 year based on population-level data for the specified disease site and stage.
* Participants with any other major medical illnesses or psychiatric treatments that in the treating physician's opinion will prevent administration or completion of protocol therapy.
* Participants with inadequate mental capacity to provide informed consent
* Participants who cannot receive gadolinium
* Participants who have undergone prior head and neck or cranial radiation or radiation to any other site previously that would be reasonably anticipated to result in a significant overlap in radiation fields.
* Participants who have received systemic or radiosensitizing therapy for a prior head and neck or central nervous system malignancy or any investigational cancer drug for glioblastoma prior to randomization.
* Participants who have received or plan to receive any other form of non-surgical local or field treatment overlapping with the anticipated radiation field.
* Patients with a serious active infection (such as a wound infection requiring parenteral antibiotics) or other acute medical conditions at the time of randomization that would impair the ability of the patient to receive protocol treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Overall survival from time of enrollment through study completion, an average of 1 year
  through study completion, an average of 1 year

SECONDARY OUTCOMES:
Progression-free survival | Time of enrollment to time of progressionfrom time of enrollment through study completion, an average of 6 months
Treatment-related toxicity | Time of enrollment to end of treatment (upto 6 months after completion of radiation therapy)
  Per CTCAE 5.0
Health-related quality of life | From time of enrollment upto 6 months later
  This will be measured by EORTC QLQ-C30 and QLQ-BN20 tools. Evaluation for changes in health-related quality of life by these instruments upto 6 months after radiation therapy.
Mood symptoms | From time of enrollment upto 6 months later
  Measured by the Patient Health Questionnaire (PHQ-4). Evaluation of changes to PHQ-4 scores over time upto 6 months after radiation treatment.
Practical Geriatric Assessment | From time of enrollment upto 6 months later
Performance status | From time of enrollment upto 6 months later
  Measured by Karnofsky Performance Status. Evaluation of changes of performance status over time upto 6 months after radiation treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Brigham Cancer Center, Milford Hospital, Milford, Massachusetts
  - Dana-Farber Brigham Cancer Center, South Shore Hospital, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
We will plan to share IPD pending securing funding to facilitate data-sharing